CLINICAL TRIAL: NCT03858244
Title: Curve Progression in Children and Adolescent Idiopathic Scoliosis With and Without Sleep-disordered Breathing
Brief Title: Idiopathic Scoliosis Progression and Sleep-disordered Breathing in Children
Status: Active, not recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: The Children's Hospital of Zhejiang University School of Medicine (Other); Ningbo No. 1 Hospital (Other); Ningbo No.2 Hospital (Other); The Third Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Xiangyang Wang, M.D., Chief physician, Doctorial supervisor, Second Affiliated Hospital of Wenzhou Medical University
Other Study IDs: SAHoWMU-CR2018-08-222
Record Dates: First submitted 2019-02-24; First posted 2019-02-28 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Scoliosis Idiopathic; Sleep Disordered Breathing; Obstructive Sleep Apnea
Keywords: Sleep; Scoliosis
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IS with SDB: Idiopathic scoliosis with untreated and treated sleep-disordered breathing
- IS without SDB, controls: Idiopathic scoliosis without sleep-disordered breathing, control group

SUMMARY:
This study aimed to investigate the prevalence and clinical significance of sleep-disordered breathing (SDB) in children with new onset and progressive idiopathic scoliosis (IS)

DETAILED DESCRIPTION:
Idiopathic scoliosis (IS) is the most common pediatric musculoskeletal disorder that causes a three-dimensional spinal deformity affecting 2 to 4% of adolescent subjects. It can be progressive (in 3 out of 10 cases) and severe involving serious effects (spine pain, cardiopulmonary compromise, deformed torso, psychosocial issues) and heavy treatments (corset, surgery). However, there is still no reliable criteria to predict the occurrence and progression of IS, while the etiology of IS remains unclear.

Sleep-disordered breathing (SDB) in children is a common condition characterized by recurrent events of upper airway obstruction during sleep. The major symptom is snoring or noisy breathing. Preliminary evidence suggests that SDB in children is associated with low bone mass and postural stability, which might be mechanisms in the development of scoliosis. However, the influence of SDB on the onset or progression of IS remains unknown.

To fill those gaps, investigators will perform a prospective, unrandomized, observational cohort study at a scoliosis center to determine the prevalence and significance of SDB in children with mild-moderate IS. All subjects will be screened with a designated sleep questionnaire (PSQ), and children with either severe daytime sleepiness or frequent snoring or any degree of sleep pause will be requested to undergo further evaluation and an overnight polysomnography (PSG). Routine follow-up visits will be scheduled 6 months apart up to at least 36 months to assess the curve progression of pre-existing scoliosis. At the same time, children with suspected curves but excluded from scoliosis at their first clinic visit will also undergo a sleep evaluation, and be uniformly screened for the new onset scoliosis in Zhejiang Province during 2023-2024. All primary and secondary school students receive annual scoliosis screening led by the Zhejiang provincial government from 2023.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic scoliosis at their first clinic visit
* Skeletally immature (Risser Sign 0-3)
* Cobb angle between 11-40 degrees
* Age between 6 and 15
* Patients can understand and complete the revised Pediatric Sleep Questionnaire at baseline and follow-up visits
* Patients with symptoms suspicious of SDB agree to undergo clinical evaluation and an overnight polysomnogram
* Informed Consent Form signed by subject or the guardian

Exclusion Criteria:

* Patients with scoliosis other than idiopathic, or with other musculoskeletal or neurodevelopmental conditions that might be responsible for the scoliosis
* History of previous spine surgery or spinal injury
* Tumor or malignant tumor in the spine
* Leg length discrepancy more than 20 mm
* Previous diagnosis or treatment of SDB more than 6 months ago
* Fail to fulfill the questionnaire or refuse to attend any further evaluation
* Severe obstructive sleep apnea syndrome (OSAS) or significant hypoxemia requiring Continuous Positive Airway Pressure treatment
* A guardian who cannot accompany the child on the night of PSG
* Plans to relocate within the next 24 months

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents with suspected or known idiopathic scoliosis that were referred to the Second Affiliated Hospital of Wenzhou Medical University
Sampling Method: Non-Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Scoliosis Curve Angle | Routine follow-up visits will be scheduled 6 months apart up to 36 months
  A long standard standing whole spine radiograph will be used for measuring curve size in terms of Cobb angle according to the standard Cobb method
Angle of Trunk Rotation | Routine follow-up visits will be scheduled 6 months apart up to 36 months
  In addition to spinal x-rays, a Scoliometer can also help monitor curve progression. The Scoliometer is an inclinometer that measures the asymmetries between the sides of the trunk by measuring axial rotation in degrees. Numerous studies have found a high correlation between trunk axial rotation (ATR) values and the Cobb angles.

SECONDARY OUTCOMES:
Sleep Measurements | Routine follow-up visits will be scheduled 6 months apart up to 36 months
  Sleep questionnaire with or without further PSG evaluation
Body mass index | Routine follow-up visits will be scheduled 6 months apart up to 36 months
  Changes in height, weight and body mass index

CONTACTS AND LOCATIONS:
Overall Officials: Xiangyang Wang, MD, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China